CLINICAL TRIAL: NCT04948606
Title: A Prospective, Observational Study Evaluating Persistence on Treatment, Safety, Tolerability, and Effectiveness of Diroximel Fumarate in the Real-World Setting (EXPERIENCE-CA+IL Study)
Brief Title: Exploring Diroximel Fumarate Real-world Experience in Canada and Israel
Acronym: EXPER-CA/IL
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-VUM-11892
Record Dates: First submitted 2021-06-28; First posted 2021-07-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Relapsing Forms of MS
Keywords: Clinically isolated syndrome; Multiple Sclerosis; Relapsing forms of Multiple Sclerosis; Active secondary progressive disease
MeSH Terms: conditions — Multiple Sclerosis | interventions — diroximel fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diroximel Fumarate (DRF): Participants with a confirmed diagnosis of MS who are newly prescribed DRF in routine clinical practice and who satisfy the approved therapeutic indication for DRF will be enrolled.
  Interventions: Drug: Diroximel Fumarate

INTERVENTIONS:
Drug: Diroximel Fumarate — Administered as specified in the treatment arm.
  Other Names: VUMERITY; BIIB098

SUMMARY:
The primary objective of the study is to characterize the persistence to therapy in participants with relapsing forms of multiple sclerosis (RMS) treated with diroximel fumarate (DRF) in routine clinical practice. The secondary objectives of the study are to assess short-term persistence to treatment; to assess long-term persistence on treatment; to assess the effect of DRF on relapses; to assess the impact of DRF on cognition; to assess the impact of DRF on participant reported outcomes (PROs); to assess the impact of DRF on disability; to assess treatment satisfaction with DRF; to explore the real-world safety profile of DRF (i.e., gastrointestinal [GI] tolerability, lymphocyte dynamics, adverse events [AEs] leading to discontinuation, and serious adverse events [SAEs].

ELIGIBILITY:
Key Inclusion Criteria:

* Have a diagnosis of MS and satisfy the approved therapeutic indication for DRF per the prescribing information.
* DRF prescribed and planned to be initiated within 60 days of enrollment or already initiated, with enrollment occurring no more than 7 days since the first dose.

Key Exclusion Criteria:

* History of gastric bypass or required use of feeding tubes.
* Current enrollment in any interventional study or in any study which may conflict with this study, per the discretion of the principal investigator (PI) and Biogen
* Have received prior treatment with DRF (more than 7 days before enrollment).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with RMS that have been prescribed DRF under standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants on Treatment with DRF | Year 1

SECONDARY OUTCOMES:
Percentage of Participants on Treatment with DRF | Month 3
Percentage of Participants on Treatment with DRF | Year 2
Annualized Relapse Rate (ARR) with DRF | Year 1 and 2
  For ARR at 1 year, the total number of days on study will be defined as the number of days since date of first dose to 1 year (365 days) if participant stay on DRF treatment for longer than 1 year, or the date of first dose to the date of DRF discontinuation if participant die or withdraw from the study prior to 1 year. For ARR at 2 years, the total number of days on study is defined as the number of days since the date of first dose to the date of DRF discontinuation. The relapse rate will be calculated as the total number of relapses experienced divided by the total number of days on DRF treatment, and the ratio multiplied by 365.
Percentage of Participants Relapsed | Year 1 and 2
Change in Cognitive Processing Speed Test (CPST) Score | Baseline, Year 1 and 2
  Change in CPST will be assessed using the Konectom application. Cognitive function will be evaluated based on elements of attention, psychomotor speed, visual processing and working memory. Cognitive function is assessed by having the participant pair abstract symbols with specific numbers using a key as a guide. Higher number of correct responses indicates better cognition
Change in Score for Each Domain of Quality of Life in Neurological Disorders (Neuro- QoL™) Questionnaire | Baseline, Year 1 and 2
  Neuro-QoL uses a T score which has a mean of 50 and SD of 10, based on the norming sample used. All Neuro-QOL banks and scales are scored such that a high score reflects more of what is being measured.
Change in Disability, as Measured by Expanded Disability Status Scale (EDSS) | Baseline, Year 1 and 2
  The EDSS measures disability status on a scale ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]), with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Mean Change in Treatment Satisfaction Questionnaire for Medication (TSQM) Score | Baseline, Year 1 and 2
  TSQM Version 1.4 is comprised of 14 questions that provide scores on four scales: effectiveness (3 items), side effects (5 items), convenience (3 items) and global satisfaction (3 items). The scale scores are transformed and range from 0 to 100. Higher scores indicate greater satisfaction.
Number of Participants with Gastrointestinal (GI) Adverse Events (AEs) | Up to Month 32
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants with AEs Leading to Treatment Discontinuation | Up to Month 32
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants with Serious Adverse Events (SAEs) | Up to Month 32
  An SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.
Number of Participants with Relevant Concomitant Medication Use | Up to Month 32
  The concomitant medication may include GI symptom medication, coronavirus disease of 2019 (COVID-19) vaccine, etc.
Number of Participants Categorized by the Types of Actions Taken Due to GI AEs | Up to Month 32
  The actions taken will include temporary dose reduction, temporary dose interruption, initiation of concomitant GI medication, taking DRF dose with food, permanent discontinuation, or other action.
Median Absolute Lymphocyte Count (ALC) Over Time | Baseline, Month 6, Year 1 and 2
Percent Change from Baseline in Median ALC | Baseline, Month 6, Year 1 and 2
Number of Participants with Lymphopenia According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI/CTCAE) Severity Grading | Up to Month 32

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (6):
- Israel (6):
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/